CLINICAL TRIAL: NCT07278180
Title: Assessment of the Effects of Platelet and Leukocyte-rich Fibrin on Vestibular Bone Plate Thickness on Alveolar Ridge Maintenance Through Three-dimensional Analysis
Brief Title: Effects of Platelet and Leukocyte-rich Fibrin on Alveolar Ridge Maintenance Through Three-dimensional Analysis
Status: Completed | Type: Observational
Sponsor: University of Guarulhos (Other)
Responsible Party: Principal Investigator, Jamil awad shibli, Investigator, University of Guarulhos
Other Study IDs: UnG 17917313.7.0000.5506
Record Dates: First submitted 2025-11-29; First posted 2025-12-11 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Caries Active; Tooth Decay; Tooth Loss / Rehabilitation
Keywords: tooth loss; decay; caries; biomaterials
MeSH Terms: conditions — Dental Caries; Tooth Loss | interventions — Transplantation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- platelet rich firbrin
  Interventions: Procedure: Alveolar socket preservation with graft and flap surgery

INTERVENTIONS:
Procedure: Alveolar socket preservation with graft and flap surgery — teeth to either the control group (coagulant-filled alveoli) or the test group (alveoli filled with platelet-rich fibrin and LPRF leukocytes)

SUMMARY:
Understanding, through accurate and reliable volumetric analysis, how the biomaterial (LPRF) and the thickness of the vestibular bone plate influence changes in bone volume after extraction, is essential for making clinical decisions that impact implant-supported rehabilitation.

ELIGIBILITY:
This prospective clinical study was conducted in accordance with the ethical principles outlined in the Declaration of Helsinki and received approval from the Research Ethics Committee of Guarulhos University, São Paulo, Brazil (CEP-UnG #. 515.153). Thirty-nine patients (24 women and 15 men), aged between 22 and 80 years, who were in overall good health, non-diabetic, periodontally healthy, non-smokers, free of blood dyscrasias, not pregnant or lactating, and requiring extraction of non-contiguous, compromised teeth due to root fractures, caries, unsuccessful endodontic treatment, root resorption, or orthodontic reasons, were enrolled.

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Subjects with indication of tooth extraction
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2016-01-20 (Actual); Primary Completion 2018-02-20 (Actual); Study Completion 2022-01-20 (Actual)

PRIMARY OUTCOMES:
bone volume after 16 weeks | 16 weeks
aveolar bone contraction | 4 months

IPD SHARING:
Plan to Share IPD: Undecided